CLINICAL TRIAL: NCT02255539
Title: Bioburden and Usability Study of the Geelong Mask System
Brief Title: Bioburden and Usability Evaluation of a Nasal Prototype CPAP Mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MA110914
Record Dates: First submitted 2014-09-24; First posted 2014-10-02 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep; sleep apnea; OSA; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPAP Nasal Mask (Experimental): Geelong Prototype Mask
  Interventions: Device: Geelong Prototype Mask

INTERVENTIONS:
Device: Geelong Prototype Mask — A nasal pillows prototype mask to be trialled with a PAP therapy device for a period of 6 weeks. Participants will wear the mask in place of their current mask for the duration of the trial.

SUMMARY:
AIM AND HYPOTHESIS: The purpose of this study is to monitor the bioburden and impedance characteristics of a prototype mask system and to evaluate the usability of the mask system. The mask system will be assessed according to objective data recordings and user questionnaires. It is hypothesised that the prototype mask components will not pose a health risk (with regards to bioburden and impedance) and that the mask system will pass usability objectives to adequately deliver CPAP treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing to give written informed consent
* Participants who can read and comprehend written and spoken English
* Participants who are over 18 years of age
* Participants who have been diagnosed with OSA
* Participants who have been established on CPAP for ≥ 6 months
* Participants currently using a ResMed nasal pillows mask

Exclusion Criteria:

* Participants who are not able to provide written informed consent
* Participants who are unable to comprehend written and spoken English
* Participants who are pregnant
* Participants who are unsuitable to participate in the study in the opinion of the researcher
* Participants with a pre-existing lung disease or a condition that would predispose them to pneumothorax (e.g. COPD, lung cancer; fibrosis of the lungs; recent (< 2years) case of pneumonia or lung infection, lung injury)
* Participants who cannot participate for the duration of the trial
* Participants who are established on bi-level support therapy
* Participants who are not established on a ResMed nasal pillows mask

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Bioburden and Impedance of the prototype mask components at 6 weeks | 6 weeks
  The population of microorganisms on mask components will be measured after 6 weeks of continuous use by a participant on their PAP therapy device to assess the safe replacement interval of the component. The impedance of the mask will also be measured to assess whether the build up of microorganisms on the mask component will affect the usability and effectiveness of the mask. Bioburden and impedance testing will be conducted in a lab environment on return of the prototype mask and components.

SECONDARY OUTCOMES:
Usability ratings of the prototype mask using a visual analog scale, compared to a reference level and the participant's current mask | 6 weeks
  Participants will be asked to complete a short questionnaire at the end of each week to evaluate the general usability of the mask system. The questionnaire will include questions related to mask comfort. The participants will answer the questions using an 11-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Schindhelm, BE PhD, Principal Investigator — Graduate School of Biomedical Engineering, University of New South Wales, Sydney Australia and Applied Research, ResMed Ltd Sydney Australia
Locations (1):
- ResMed Ltd, Sydney, New South Wales, Australia